CLINICAL TRIAL: NCT04651751
Title: Facilitating an Exercise Habit and Identity Via the Multi-Process Action Control Model- A Randomized-Controlled Trial
Brief Title: Exercise Habit & MPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Victoria (Other)
Responsible Party: Principal Investigator, Ryan Rhodes, Professor, University of Victoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AT956
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Public Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No Intervention: Control Participants exercised on their own without receiving any instructions.
- Intervention (Experimental): Those who were randomized into the intervention group attended a workshop where the PI delivered a presentation that focused on establishing a preparatory exercise habit by using the M-PAC approach and proposed habit model. Participants were then provided with instructions on completing their exercise plan sheet.
  Interventions: Behavioral: Facilitating an Exercise Habit and Identity via the Multi-Process Action Control Model- A Randomized-Controlled Trial

INTERVENTIONS:
Behavioral: Facilitating an Exercise Habit and Identity via the Multi-Process Action Control Model- A Randomized-Controlled Trial — Participants attended a workshop which consisted of a presentation and an exercise planning exercise.
  Arms: Intervention

SUMMARY:
The limitations of applying social cognitive models to understand physical activity (PA) have led to the emergence of several new PA models within the past decade. The Multi-Process Action Control (M-PAC) is a comprehensive PA model that proposes intention is established from outcome expectations, perceived capability, and opportunity, then the success of translating this to behavior depends on affective judgments and behavioral-regulation. Over time, M-PAC proposes that behavior is can become maintained through the formation of identity and habit. The purpose of this study was to investigate the trajectory of change of these M-PAC constructs across time in a randomized controlled trial. Participants (n=85) were inactive new gym members and were randomized into a control (n=41) or intervention (n=44) group. The intervention group attended a workshop and received a booster phone call follow-up at week four. Measures for both groups included accelerometry and M-PAC at baseline and eight week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-65
* new gym members
* exercising < 150 minutes/week at a moderate to vigorous level

Exclusion Criteria:

* not affiliated with a gym or recreation center
* exercising > 150 minutes/week at a moderate to vigorous level
* clinical health conditions (assessed by the PAR-Q)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
GT3X+ Actigraph Activity Monitors (for measuring physical activity) | Baseline to 8 weeks
  Participants wear accelerometers for one week at baseline and at week eight to record their physical activity.

SECONDARY OUTCOMES:
1.Self-Report Behavioural Automaticity Index (self report, survey question | Baseline, week four, week eight
  The Self-Report Behavioral Automaticity Index (SRBAI) was used to assess preparatory habit. The SRBAI consists of 4 items on a 5-point Likert scale with 1 being strongly disagree to 5 being strongly agree. The question stem stated ''When I prepare to exercise…'' which was then followed by four items on the scale: ''I do it without having to consciously remember'', ''I do it automatically'', ''I do it without thinking'', and ''I start before I realize I am doing it''.

OTHER OUTCOMES:
Environmental Cues (self report, survey question) | Baseline, week four, week eight
  The following item was used to assess if participants implemented the use of cues: "I use cues at home to remind me to exercise (e.g. placing a water bottle on my desk or gym clothes on the bed). The item was rated on a five point Likert scale which ranged from "1=strongly disagree" to "5= strongly agree".
Temporal Consistency (self report, survey question) | Baseline, week four, week eight
  The item was worded "How consistently do you exercise at the same time each day? (e.g., exercising every morning at 7 am, or exercising daily after supper)". The question was asked on a five point Likert scale which range from "1=not consistent at all" to "5=very consistent".

CONTACTS AND LOCATIONS:
Overall Officials: Ryan E Rhodes, PhD, Study Chair — University of Victoria